CLINICAL TRIAL: NCT02472314
Title: A Novel Application of Exparel for Postoperative Pain Management in Shoulder Arthroplasty and Humerus Fracture Fixation
Brief Title: Exparel for Postoperative Pain Management in Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Vani J. Sabesan, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-193
Record Dates: First submitted 2015-06-03; First posted 2015-06-15 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Fracture of Shoulder and Upper Arm
MeSH Terms: conditions — Shoulder Fractures | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Liposomal Bupivacaine A (Experimental): One time injection of 1.3% Liposomal Bupivacaine during shoulder arthroplasty
  Interventions: Drug: 1.3% Liposomal Bupivacaine
- CISB control for A (Active Comparator): Peripheral nerve block (CISB) with 0.125% bupivacaine during shoulder arthroplasty .
  Interventions: Drug: 0.125% Bupivacaine
- Liposomal Bupivacaine B (Experimental): One time injection of 1.3% Liposomal Bupivacaine during Humerus Fracture Fixation
  Interventions: Drug: 1.3% Liposomal Bupivacaine
- CISB control for B (Active Comparator): Peripheral nerve block (CISB) with 0.125% bupivacaine during fracture fixation
  Interventions: Drug: 0.125% Bupivacaine

INTERVENTIONS:
Drug: 1.3% Liposomal Bupivacaine — local tissue infiltration of Liposomal Bupivacaine during surgery
  Other Names: Exparel
  Arms: Liposomal Bupivacaine A; Liposomal Bupivacaine B
Drug: 0.125% Bupivacaine — Continues nerve block with Bupivacaine during surgery and postoperatively
  Other Names: Bupivacaine
  Arms: CISB control for A; CISB control for B

SUMMARY:
The purpose of this study is to compare the effect of liposomal Bupivacaine infiltration into the shoulder to continues nerve block with Bupivacaine on postoperative pain control and functional outcomes.

DETAILED DESCRIPTION:
liposomal bupivacaine analgesia will provide improved postoperative pain control, reduction in amount of opioid supplementation, decreased complications and faster return to function compared to current standard of care pain management for patients undergoing shoulder arthroplasty and shoulder surgery for proximal humerus fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing shoulder arthroplasty under general anesthesia
* Patients undergoing open reduction internal fixation (ORIF) of a proximal humerus fracture under general anesthesia
* Patients with American Society of Anesthesiologist (ASA) physical status classification of 1-3
* Patients meeting criteria for standard of care continuous peripheral nerve block (CPNB) per anesthesia guidelines.
* Patients agreeing to be available for brief follow up telephone survey post- operatively and being mentally able to respond.
* Patients available for follow up routine post-operative clinic visits, per standard of care.

Exclusion Criteria:

* Contraindications to regional anesthesia
* Significant peripheral neuropathy or neurological disorder affecting the upper extremity
* Contraindication to a component of multimodal analgesia
* Pregnancy
* Opioid tolerance
* Cognitive or psychiatric condition that might affect patient assessment and/or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University Physician Group, Dearborn, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, randomized, controlled study included 70 consecutive shoulder arthroplasty patients from August 2015 through June 2016 during the period of 1 year at one location.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
Started | 34 | 36
Completed | 34 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine A | CISB Control for A | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 36 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 25 | 19 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 36 | 70
Surgical Side [Count of Participants; unit: Participants]
  Left | 18 | 17 | 35
  Right | 16 | 19 | 35
Arthroplasty type [Number; unit: participants]
  Hemi | 1 | 1 | 2
  Reverse | 16 | 20 | 36
  Total | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Quality of Analgesia
Description: Quality of analgesia as measured by numerical rating scores for pain (active and at rest) as (0=no pain, 10= worst pain) every two hours for the initial 36 hours, then on day2, day7 and day30 postoperatively
Time Frame: 30 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
Number analyzed (Participants) | 34 | 36
score on a scale
  At 24 to 48 hours | 2.1 [0 to 10] | 2.6 [0 to 10]
  Day 2 | 4.1 [0 to 10] | 4.0 [0 to 10]
  Day 7 | 3.4 [0 to 10] | 2.6 [0 to 10]
  Day 30 | 2.0 [0 to 10] | 2.2 [0 to 10]

2. Secondary Outcome: Post Operative American Shoulder and Elbow Surgeons (ASES)
Description: American Shoulder and Elbow Surgeons (ASES) score is an outcome reporting measure for assessments of shoulder function in patients with shoulder pathology and after shoulder arthroplasty surgery. ASES is a 100 points scale consisting of two measures: one pain scale (worth 50 points) and 10 activities of daily living(worth 50 points), the total score is the sum of both and the higher total score indicates better outcome.
Time Frame: Preoperative, 6 weeks and last follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
Number analyzed (Participants) | 34 | 36
score on a scale
  Pre-operative | 36.1 (20.04) | 27.7 (15.7)
  6 Weeks after surgery | 59.5 (18.1) | 57.3 (16.2)
  Last Followup | 74.5 (22.7) | 59.7 (20.5)

3. Secondary Outcome: Subjective Shoulder Value (SSV)
Description: Functional assessments after shoulder arthroplasty surgery. The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%. The range is between 0% and 100%
Time Frame: Pre-operative, 6 weeks and last Follow up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
Number analyzed (Participants) | 34 | 36
score on a scale
  Preoperative | 30.7 [0 to 100] | 24.3 [0 to 100]
  at 6 weeks post-op | 55.7 [0 to 100] | 63.1 [0 to 100]
  At last follow up | 70.0 [0 to 100] | 69.3 [0 to 100]

4. Secondary Outcome: Incidence of Nerve Injury
Description: Neuropraxia on the treatment side
Time Frame: During hospital stay and at 2 weeks and 6 weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
Number analyzed (Participants) | 34 | 36
Participants | 0 | 0

5. Secondary Outcome: Post Operative Opioid Consumption
Description: Cumulative amount of opioids administered during the time frame
Time Frame: During hospital stay up to 48 hours after surgery
Measure: Number; unit: Total MME per Group
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
Number analyzed (Participants) | 34 | 36
Total MME per Group | 78.6 | 52.8

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Liposomal Bupivacaine A | CISB Control for A
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/36
Other Adverse Events (participants affected / at risk) | 1/34 | 7/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine A (N=34) | CISB Control for A (N=36)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Respiratory insufficiency in a chronic obstructive pulmonary disease and sleep apnea
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine A (N=34) | CISB Control for A (N=36)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
catheter malposition (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Residual numbness of the hand and neck
Catheter fall out (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
* The NRS pain scale has been associated with higher patient-reported pain scores
* Surgeons were not blinded to intervention as they had to perform the injection
* Surgeons were involved with the assessment portion of the outcome evaluations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT02472314/Prot_SAP_000.pdf